CLINICAL TRIAL: NCT01517633
Title: Study of a Diagnostic Device for Identifying Between Amniotic Fluid to Urine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300165-HMO-CTIL
Record Dates: First submitted 2012-01-23; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Amniotic Fluid Leakage
Keywords: Amniotic fluid leakage; Urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

ARMS (1):
- A device for identifying between amniotic fluid and urine (Experimental)
  Interventions: Device: BirthSign

INTERVENTIONS:
Device: BirthSign — When leakage from the vagina occurs, the woman will wet the indicator lines of the device with the body fluids.

SUMMARY:
The purpose of this study is to compare the reliability and validity of a new device with standard methods for diagnosing between amniotic fluid leakage due to premature rupture of the membranes (PROM) and urine.

DETAILED DESCRIPTION:
Pregnant women sensing wetness and arriving to the delivery room with suspect PROM will use a self-testing device to test whether the wetness is caused by amniotic fluid leakage or urinary incontinence. Clinical evaluation will be performed to all pregnant women using standard clinical tests. The results of the standard clinical tests will be compared to the women's reading of the self-testing device results. Sensitivity and specificity of the device evaluation will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women age 18 years and older attending delivery room.
2. Stage of gestation: pregnancy between 16 and 42 weeks of gestation.
3. Able and willing to read and sign an informed consent document.

Exclusion Criteria:

Subjects will be excluded from the study if any of the following will be present:

1. Prior use of any amniotic fluid detection test.
2. Use of vaginal douching apparatus (such as a vaginal bulb syringe) or vaginal products such as creams or gels within the past 24 hours.
3. Vaginal bleeding or spotting or excess abnormal vaginal discharge within the past 24 hours.
4. Sexual intercourse within the past 24 hours.
5. Confirmed diagnosis of any vaginal infection within the past 7 days.
6. Use of vaginal products or antibiotic treatments that reduce bacterial population or use of medications such as tamoxifen that reduce estrogen levels or antihistamines that dry mucous membranes within the past 7 days..
7. Patients unable or unwilling to participate.
8. Patients in active labor (or with regular contractions).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Presence / absence of stains comparing to a known color index printed on the product | 12 hours
  Presence / absence of a blue-green stain and / or brown-red stain as yielded by the device and observed by the woman.

SECONDARY OUTCOMES:
Presence / absence of stains comparing to a known color index printed on the product | 12 hours
  Presence / absence of a blue-green stain and / or brown-red stain as yielded by the device and observed by the clinician and a measurement of patient comfort while using the device, reading the results and clarity of instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] El-Messidi A, Cameron A. Diagnosis of premature rupture of membranes: inspiration from the past and insights for the future. J Obstet Gynaecol Can. 2010 Jun;32(6):561-569. doi: 10.1016/S1701-2163(16)34525-X. PMID 20569537